CLINICAL TRIAL: NCT01092559
Title: An Open Label Pilot Study Evaluating Preliminary Safety and Performance of the GeNO Nitrosyl Delivery System
Brief Title: Pilot Study Evaluating the Safety and Performance of the GeNO NITROsyl Delivery System for Inhaled Nitric Oxide
Acronym: PILOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geno LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P2010-001
Record Dates: First submitted 2010-02-16; First posted 2010-03-25 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Diagnostic Techniques and Procedures
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nitric oxide via GeNO Nitrosyl system (Experimental): Nitric Oxide via GeNO Nitrosyl system
  Interventions: Drug: Nitric Oxide generated by the GeNO nitrosyl delivery system

INTERVENTIONS:
Drug: Nitric Oxide generated by the GeNO nitrosyl delivery system — single short-term exposure to inhaled nitric oxide using the GeNO nitrosyl delivery system.

SUMMARY:
This is an open label phase 2 pilot study designed to evaluate the safety, tolerability and device performance of the GeNO nitrosyl delivery system during right heart catheterization (RHC) in participants with pulmonary arterial hypertension (PAH). All participants will receive inhaled nitric oxide in oxygen or nitric oxide in air delivered by nasal cannula. Hemodynamics, clinical laboratory and clinical assessment data will be collected on all participants to evaluate safety.

DETAILED DESCRIPTION:
TREATMENT/FOLLOW-UP:

Participants meeting eligibility criteria will receive open label nitric oxide at 80 ppm via a nasal cannula. Hemodynamic clinical laboratory and clinical assessment data will be collected at baseline, after 15 minutes of inhaled nitric oxide administration, post RHC procedure and at hospital discharge. Day 5 +/- 3 post RHC, telephone contact to assess general health status.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of PAH, WHO Group 1.
* WHO Functional Class II or III equivalent, PAH.
* Have been clinically stable with regard to signs and symptoms of PAH for at least 30 days prior to RHC.
* May be receiving approved mono therapies or combination PAH therapies.
* Females that are surgically sterile or post-menopausal. Females of chil-bearing potential must have negative pregnancy test and must be practicing adequate birth control.

Exclusion Criteria:

* Have had a new type of chronic therapy (including but not limited to oxygen, a different category of vasodilator, a diuretic, digoxin) for PAH added within (1) month of RHC.
* Have any PAH medication except for anticoagulants discontinued within the week prior to RHC.
* Have evidence of significant parenchymal lung disease as evidenced by pulmonary function tests within the last six months
* CREST (calcinosis, Raynaud phenomenon, esophageal dysmotility, sclerodactyly, telangiectasia) syndrome
* Have a history of uncontrolled sleep apnea within three months of RHC.
* Have a history of hemodynamically significant left-sided heart disease
* Have evidence of left-sided heart disease
* Have any other disease that is associated with pulmonary hypertension (e.g. congenital systemic-to-pulmonary shunt, sickle cell anemia, schistosomiasis).
* Documented uncontrolled systemic hypertension as evidenced by systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg.
* Have used prescription appetite suppressants within 3 months prior to wean/transition.
* Have chronic kidney disease stage IV or worse or the requirement for dialysis.
* Be receiving an investigational drug, have in place an investigational device, or have participated in an investigational drug study within the past 30 days.
* Have had an atrial septostomy.
* Have anemia (hemoglobin <10 g/dL), active infection or any other ongoing condition that would interfere with the interpretation of study assessments.
* Have any serious or life-threatening disease other than conditions associated with PAH (e.g. malignancy requiring aggressive chemotherapy, renal dialysis, etc.).
* Have unstable psychiatric status or be mentally incapable of understanding the objectives, nature or consequences of the trial
* Participant is pregnant or lactating
* Significant, ongoing alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tufts, Boston, Massachusetts
  - University Hospital, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitric Oxide Via GeNO Nitrosyl System: Nitric Oxide generated by the GeNO nitrosyl delivery system : single short-term exposure to inhaled nitric oxide using the GeNO nitrosyl delivery system.
Period: Overall Study
Arm/Group | Nitric Oxide Via GeNO Nitrosyl System
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nitric Oxide Via GeNO Nitrosyl System
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (15.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment Emergent Adverse Events; Unanticipated Adverse Device Effects and Changes From Baseline to End-of-study in Clinical Lab Parameters and Vital Signs.
Description: Adverse Event Severity [through Day 30 Follow-Up Period]
  Unanticipated Device Effects: any system malfunction, damage or NO2 threshold monitor alarms [through discharge from Treatment Period]
  Laboratory Tests: Hematology (CBC with differential), Chemistry (glucose, BUN, creatinine, sodium, potassium, carbon dioxide, creatinine kinase), Activated Clotting Test or Prothrombin Time, arterial blood gas, and methemoglobin.
  [through discharge from Treatment Period]
  Vital Signs: pulse, blood pressure, respiratory rate [through discharge from Treatment Period]
Time Frame: through Day 30 Follow-up Period
Measure: Number; unit: participants
Arm/Group | Nitric Oxide Via GeNO Nitrosyl System
Number analyzed (Participants) | 10
participants | 0

2. Primary Outcome: Adequacy of Device Design and Suitability of the Instructions for Use by the Clinician Using a Device Performance Evaluation
Time Frame: through Treatment Period
Measure: Number; unit: participants
Arm/Group | Nitric Oxide Via GeNO Nitrosyl System
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Arm/Group | Nitric Oxide Via GeNO Nitrosyl System
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less